CLINICAL TRIAL: NCT06970873
Title: Evaluation of Knowledge, Attitude, and Practice of Pediatric Dentists Toward Obstructive Sleep Apnea Among Children in Egypt: A Cross-sectional Study
Brief Title: Knowledge, Attitude, and Practice of Pediatric Dentists Toward Obstructive Sleep Apnea Among Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Aly, Associate professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 22-2-25
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Knowledge; Attitude; practice; Pediatric Dentist; Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric dentists
  Interventions: Other: Evaluation of Knowledge, Attitude, and Practice of Pediatric Dentists

INTERVENTIONS:
Other: Evaluation of Knowledge, Attitude, and Practice of Pediatric Dentists — Evaluation of Knowledge, Attitude, and Practice of pediatric dentists toward Obstructive Sleep Apnea among Children

SUMMARY:
The main objective of this study is to assess the knowledge, attitude, and practice of Egyptian pediatric dentists toward obstructive sleep apnea among children.

DETAILED DESCRIPTION:
Data will be collected using a self-administrated questionnaire developed based on a previous study. The questionnaire was delivered to pediatric dentists, including both dental faculty and practitioners specializing in pediatric dentistry through E-mail and administered in the English language using the Google Forms platform.

The questionnaire began with an invitation message, followed by a consent agreement for participation. It was divided into four sections: demographic information, knowledge about obstructive sleep apnea, attitude toward obstructive sleep apnea, and practice related to obstructive sleep apnea. The demographic section collected information on respondents' age, gender, practice sector (primary health center or private clinic), and years of experience.

The knowledge section comprised questions based on the definition of obstructive sleep apnea, followed by 17 knowledge statements to assess the extent of dentists' knowledge about obstructive sleep apnea. These statements covered topics such as prevalence, percentage of affected individuals, symptoms, diagnosis, risk factors, treatment, and the role of dentists in managing obstructive sleep apnea. Response options included "true," "false," and "do not know." Correct answers were awarded 1 point, whereas incorrect answers received no points. The inclusion of the "do not know" option aimed to minimize guessing and was scored as an incorrect response.

The attitude section consisted of seven questions focusing on the role of pediatric dentists in diagnosing and treating obstructive sleep apnea in children, screening for obstructive sleep apnea based on snoring history, considering obstructive sleep apnea screening as a mandatory part of clinical examination, and the need to include obstructive sleep apnea information in the undergraduate curriculum. The response scale for the attitude section included "yes" (1 point awarded, indicating a positive attitude) or "no" or "do not know" (no points awarded, indicating a negative attitude).

The practice section encompassed five questions, exploring whether pediatric dentists had fabricated oral appliances for managing obstructive sleep apnea, their approach to history taking including questions to rule out the presence of obstructive sleep apnea, and their participation in continuing education courses related to the topic.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric dentists

Exclusion Criteria:

* Undergraduate student

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric dentists
Sampling Method: Probability Sample
Enrollment: 362 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Pediatric Dentists toward Obstructive Sleep Apnea among Children | 1 month
  Knowledge of Pediatric Dentists toward Obstructive Sleep Apnea among Children measured by questionnaire with close ended questions

SECONDARY OUTCOMES:
Attitude of Pediatric Dentists toward Obstructive Sleep Apnea among Children | 1 month
  Attitude of Pediatric Dentists toward Obstructive Sleep Apnea among Children measured by questionnaire using close ended questions
Practice of Pediatric Dentists toward Obstructive Sleep Apnea among Children | 1 month
  Practice of Pediatric Dentists toward Obstructive Sleep Apnea among Children using questionnaire composed of close ended questions

REFERENCES:
- [Derived] Aly MM, Elchaghaby MA, Yousry YM. Pediatric obstructive sleep apnea: knowledge, attitude, and practice among pediatric dentists in Egypt: a cross-sectional study. BMC Oral Health. 2025 Sep 23;25(1):1417. doi: 10.1186/s12903-025-06944-w. PMID 40988011